CLINICAL TRIAL: NCT06777017
Title: Can Hepatic-splenic Elastography Predict the Risk of Hepatocellular Recurrence After Radiofrequency Ablation?
Acronym: ELASTORFA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ELASTORFA
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to assess whether there is an association between hepatic and splenic elastography values and the risk of HCC recurrence after treatment with RFA

DETAILED DESCRIPTION:
The primary objective of the study will be to assess whether there is an association between hepatic and splenic elastography values and the risk of HCC recurrence after treatment with RFA. Secondary objectives, however, will be to test whether hepatic and splenic elastography values have an association with overall and HCC-related survival and with the risk of decompensation after treatment with RFA; further secondary objective will be to evaluate the association between non-invasive biochemical tests and the risk of HCC recurrence after treatment with RFA. The population will consist of hepatopathic patients with HCC who are candidates for treatment with RFA and who are referred to the coordinating center "U.O.C. of Gastroenterology and Digestive Endoscopy" of IRCSS Azienda Ospedaliero-Universitaria, Policlinico di S.Orsola and the Participating Center "U.O. of Gastroenterology," Azienda Ospedaliero-Universitaria Integrata di Modena.

ELIGIBILITY:
Inclusion Criteria:

* Clinical-instrumental diagnosis of chronic liver disease.
* Indication for treatment of HCC with RFA using the Barcelona Clinic Liver Cancer (BCLC staging system) classification system19;
* Performing hepatic or splenic elastography by transient method with Fibroscan® (Echosens, Paris, France) or ARFI method (ACUSON Sequoia Siemens).
* Signature of informed consent

Exclusion Criteria:

* Age < 18 years;
* Diagnosis of hepatocholangiocarcinoma or other hepatic focal lesions other than hepatocellular carcinoma;
* Previous history of liver transplantation (OLT) and/or liver resection for HCC in the previous two years;
* Liver disease in decompensation (Child-Pugh C) at the time of informed consent or within three months prior to enrollment;
* Patients with other severe and advanced diseases that may affect short-term mortality (e.g. further non-remission neoplasms, heart failure >NYHA III, chronic renal failure in dialysis, pulmonary diseases dependent on home oxygen therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hepatopathic patients with HCC who are candidates for treatment with RFA and who are admitted to the coordinating center "U.O.C. of Gastroenterology and Digestive Endoscopy" of the IRCSS University Hospital Company, Policlinico di S.Orsola and to the Participating Center "U.O. of Gastroenterology", Integrated University Hospital of Modena are eligible to enter the study. Patients who meet the inclusion criteria will be enrolled in the study. Patients may be enrolled during treatment-preventive outpatient visits, during the elastographic examination or at the time of scheduled admission to the participating U.O. for the execution of the treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between hepatic and splenic elastography values and the risk of HCC recurrence after treatment with RFA | 12 months
  The primary objective of the study will be to assess whether there is an association between hepatic and splenic elastography values and the risk of HCC recurrence after treatment with RFA

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Maurizio Zagari, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, Bologna, Italy